CLINICAL TRIAL: NCT05031949
Title: A Single-center, Single-arm, Non-randomized Clinical Study to Evaluate the Efficacy and Safety of Hyperbaric Oxygen Therapy Plus Camrelizumab as a Second-line Treatment in Advanced/Metastatic Hepatocellular Carcinoma
Brief Title: Hyperbaric Oxygen Therapy Combined Camrelizumab in Patients With Advanced/Metastatic Hepatocellular Carcinoma
Acronym: CCGLC-003
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhang Bi Xiang, MD (Other)
Responsible Party: Sponsor-Investigator, Zhang Bi Xiang, MD, Prof.; M. D.; Ph. D., Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-S087
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Combinational Immunotherapy; Hepatocellular Carcinoma Non-Resectable; Hyperbaric Oxygen Therapy
Keywords: hyperbaric oxygen therapy; Camrelizumab; hepatocellular carcinoma; second-line treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hyperbaric Oxygenation; camrelizumab

STUDY DESIGN:
Intervention Model Description: A Phase 1b, Open-Label, Single-Arm Study to explore the efficacy and safety of hyperbaric oxygen therapy plus Camrelizumab as a second-line treatment in patients with advanced hepatocellular carcinoma who have failed at least 1 previous treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperbaric oxygen therapy plus Camrelizumab (Experimental): Subjects receive Camrelizumab intravenous at the dose 3mg/kg on Day 1 every 3 weeks, and breath pressurized (0.25 MPa) 100% oxygen (O2) indirectly by a head hood or mask for 60 minutes in multiplace chambers at Day 1 of every week.
  Interventions: Combination Product: hyperbaric oxygen therapy plus Camrelizumab

INTERVENTIONS:
Combination Product: hyperbaric oxygen therapy plus Camrelizumab — Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody

SUMMARY:
The purpose of this study is to explore the efficacy and safety of hyperbaric oxygen therapy plus Camrelizumab as a second-line treatment in patients with advanced hepatocellular carcinoma who have failed at least 1 previous treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteer to participate in the study and agree to sign the informed consent with good compliance and follow-up.
2. Subjects are 18 years old or older when signing the informed consent and gender is not limited.
3. Histologically confirmed HCC in advanced stage; not suitable to surgery or local regional treatment; with at least one measurable lesion per RECIST 1.1
4. Failed or intolerable to at least one prior systemic treatment for advanced HCC
5. With at least one assessment lesion according to the RESIST v1.1 criteria.
6. Estimated survival time ≥ 12 weeks.
7. The ECOG score is 0-1 within 1 week before enrollment.
8. Adequate organ function, including:

   1. Whole blood cell examination (no blood transfusion within 14 days, no G-CSF use and no drugs use): Hb≥90g/L, ANC≥1.5×10*9/L, PLT≥70×10*9/L;
   2. Biochemical examination (no ALB infused within 14 days): ALB≥29 g/L, ALT and AST<5×ULN, TBIL≤1.5×ULN, creatinine≤1.5×ULN, and prothrombin time or INR ≤1.5×ULN;
   3. thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
9. Without biliary obstruction. Subjects who need biliary stent implantation must be completed at least 7 days before enrollment
10. Male or female participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 60 days for female subjects and 120 days for male subjects after the last dose of study drug
11. Subjects with asymptomatic or stable brain metastases after local treatment are allowed to be included as long as they meet the following conditions:

    1. measurable lesions outside the central nervous system;
    2. No central nervous system symptoms or no aggravation of symptoms for at least 2 weeks;
    3. Those who do not need glucocorticoid treatment or stop glucocorticoid treatment within 7 days before the administration of the first study drug;
    4. Patients were allowed to receive palliative radiotherapy, but the end time of radiotherapy was within 7 days before the administration of the first study drug.

Exclusion Criteria:

Subjects with one or more than one of the following criteria should be excluded

1. Subjects has contraindications of hyperbaric oxygen use, including pneumothorax, mediastinal edema, multiple rib fractures, open trauma of chest wall, vacuolar pulmonary tuberculosis with hemoptysis, pulmonary bullae, active internal bleeding and hemorrhagic diseases;
2. Subjects with other malignant tumors in the past 5 years (radical skin basal cell carcinoma, skin squamous epithelial carcinoma, and / or radical resection of carcinoma in situ were not included);
3. subjects are currently participating in other interventional clinical studies, or received any topical treatment within 4 weeks prior to the study, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection;
4. systemic treatment with traditional Chinese medicine with anti-tumor indications or drugs with immunomodulatory effect (including thymosin, interferon and interleukin, except for local use to control pleural effusion) within 2 weeks before the first administration;
5. Diagnosis of immunodeficiency or systemic steroid therapy or any form of immunosuppressants therapy within 7 days prior to this study. A physiological dose of corticosteroids (no more than 7.5 mg/d prednisone or equivalent) can be approved after clinical evaluation;
6. Pleural effusion or Ascites with clinical symptoms which requires pleural or abdominal puncture or drainage therapy;
7. Subjects have organ transplantation history.
8. Subjects are allergic to the active ingredients or excipients of Camrelizumab;
9. Subjects with multiple factors affecting oral drugs (such as inability to swallow, post gastrointestinal resection, chronic diarrhea and intestinal obstruction);
10. Not fully recovered from toxicity and / or complications caused by any intervention before starting treatment (i.e. ≤ grade 1 or reaching baseline, excluding fatigue or hair loss);
11. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1 / 2 antibody positive);
12. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number at the same time was higher than the upper limit of normal value in the laboratory of the research center).Note: hepatitis B patients who meet the following criteria can also be enrolled:

    1. Before the first administration, the HBV viral load was less than 1000 copies / ml (200 IU / ml). Subjects should receive anti HBV treatment throughout the study chemotherapy treatment to avoid virus reactivation;
    2. For subjects with anti HBC (+), HBsAg (-), anti HBS (-) and HBV viral load (-), preventive anti HBV treatment is not required, but virus reactivation needs to be closely monitored.
13. Active HCV infected subjects (HCV antibody positive and HCV-RNA level higher than the lower limit of detection);
14. Live vaccine was administered within 30 days before the first administration (cycle 1, day 1);Note: it is allowed to receive inactivated virus vaccine for injection against seasonal influenza within 30 days before the first administration; However, live attenuated influenza vaccines administered intranasal are not allowed.
15. Female subjects who are pregnant, breastfeeding or refuse contraception.
16. Subjects have any serious or uncontrollable systemic diseases, such as:

    1. There are significant abnormalities in rhythm, conduction or morphology of resting ECG and the symptoms are serious and difficult to control, such as complete left bundle branch block, heart block above grade II, ventricular arrhythmia or atrial fibrillation;
    2. Unstable angina pectoris, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) grade ≥ 2;
    3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before enrollment;
    4. Poor blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
    5. A history of noninfectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or the current presence of clinically active interstitial lung disease;
    6. Active pulmonary tuberculosis;
    7. There are active or uncontrolled infections requiring systemic treatment;
    8. There were clinically active diverticulitis, abdominal abscess and gastrointestinal obstruction;
    9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
    10. Diabetes was poorly controlled (fasting blood glucose (FBG) > 10mmol/L).
    11. Urine routine examination showed that urinary protein was ≥ + +, and the 24-hour urinary protein was confirmed to be more than 1.0 G;
    12. Subjects with mental disorders and unable to cooperate with treatment;
17. Subjects are unsuitable for participation in this research after comprehensive assessment by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1 | up to 12 months.
  ORR defined as the proportion of subjects who achieved a complete response (disappearance of all target lesions) or a partial response (≥ 30% decrease in the sum of the longest diameters of target lesions) based on RECIST v1.1.
Progression-free survival based on RECIST v1.1 | Time from first treatment to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival defined as the time from the first day of taking study drug to death or disease progression by RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Response Rate per RECIST v1.1 | up to 12 months
  time from the date of CR or PR until PD
Disease control rate per RECIST v1.1 | up to 12 months
  Disease control rate (DCR)=CR + PR + stable disease
Overall Survival | up to 12 months
  Duration from the date of initial treatment with hyperbaric oxygen therapy plus Camrelizumab to the date of death due to any cause.
Number of Subjects with one or more adverse events as assessed by CTCAE 5.0 | From screening through 30-35 days after end of treatment, up to 12 months
  Safety and tolerability of hyperbaric oxygen therapy plus Camrelizumab as assessed by the frequency, duration, and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatic Surgery Center, Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China